CLINICAL TRIAL: NCT04632472
Title: Targeted Left Ventricular Lead Placement for Cardiac Resynchronization Therapy, a Randomized Trial Comparing an Active Fixation Bipolar Left Ventricular Lead and Passive Fixation Quadripolar Leads
Brief Title: Targeted Left Ventricular Lead Placement, Comparison of Active Fixation Bipolar and Passive Quadripolar Pacemaker Leads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1507
Record Dates: First submitted 2020-11-03; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization therapy
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient blinded The echocardiographic analyses were done blinded to type of left ventricular lead.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active fixation bipolar lead (Active Comparator): Left ventricular bipolar pacemaker lead, fixated by a side helix
  Interventions: Device: Active fixation bipolar lead versus passive fixation quadripolar leads in Cardiac Resynchronization Therapy
- Passive fixation quadripolar lead (Placebo Comparator): Left ventricular quadripolar passive fixation pacemaker lead
  Interventions: Device: Active fixation bipolar lead versus passive fixation quadripolar leads in Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Active fixation bipolar lead versus passive fixation quadripolar leads in Cardiac Resynchronization Therapy — Cardiac resynchronization therapy trial comparing types of leads.

SUMMARY:
A prospective, randomized and patient-blinded trial comparing an active fixation left ventricular lead with quadripolar passive left ventricular leads. The leads were compared in order to identify differences in the electrical performance, the ability to achieve a stable proximal position in a coronary vein located concordant to target segment and clinical outcome. The patients were followed up for 12 months.

DETAILED DESCRIPTION:
A prospective, randomized and patient-blinded trial. The objective was to compare an active fixation left ventricular lead with quadripolar passive left ventricular leads. The left ventricular segment with latest mechanical activation was identified as target segment by radial strain speckle-tracking echocardiography.The leads were compared in order to identify differences in the electrical performance, the ability to achieve a stable proximal position in a coronary vein located concordant to target segment and clinical outcome. The clinical outcomes were assessed by echocardiography, change in New York Heart Association (NYHA) functional class and Minnesota Living With Heart Failure Questionnaire (MLHFQ). The patients were followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) ≤ 35 %
* NYHA 2-4
* Electrocardiogram : left bundle branch block (LBBB) and QRS duration >120 ms or non-LBBB and QRS duration ≥150 ms
* Optimal medical treatment.

Exclusion Criteria:

* Upgrade procedures due to ventricular pacing
* No written consensus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Echocardiographic response | Day 0 (baseline). 6 and 12 months after implantation
  Changes in left ventricular end-systolic volume (measured in milliliter).
Ability to achieve a position in a coronary vein located concordant to target segment. | At implant (day 0)
  The left ventricular lead final position will be compared to the left ventricular target segment. The target segment is determined by radial strain speckle-tracking echocardiography. The lead position is classified as "concordant" or "not concordant".
The left ventricular lead long-axis position. | At implant (day 0)
  Measurement of the distance (millimeter) from the active electrode to coronary sinus. Fluoroscopic measurement in a right anterior oblique (RAO) view.
The left ventricular lead pacing threshold | Day 0 (baseline). 2, 6 and 12 months after implantation.
  Changes in left ventricular lead pacing capture thresholds, measured in "Volt" with 0.4ms pulse width.

SECONDARY OUTCOMES:
Changes in NYHA functional Class | Day 0 (baseline). 2, 6 and 12 months after implantation
  Assessment of NYHA functional Class. Class I - No symptoms and no limitation in ordinary physical activity. Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms. Class IV - Severe limitations, symptoms even while at rest.
Changes in MLHFQ score | Day 0 (baseline). 2, 6 and 12 months after implantation
  Evaluating Quality of Life. 21 questions with total scores ranging from 0 to 105. A higher score means a worse outcome.
Left ventricular lead impedances | Day 0 (baseline). 2, 6 and 12 months after implantation
  Changes in left ventricular pacing impedances, measured in "Ohm".
Changes in left ventricular ejection fraction | Day 0 (baseline). 6 and 12 months after implantation.
  Changes in left ventricular ejection fraction (unit:"percent") measured by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Department of Heart Disease, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keilegavlen H, Schuster P, Hovstad T, Faerestrand S. Clinical outcome of cardiac resynchronization therapy in patients randomized to an active fixation bipolar left ventricular lead versus a passive quadripolar lead. Scand Cardiovasc J. 2021 Jun;55(3):153-159. doi: 10.1080/14017431.2020.1869299. Epub 2021 Jan 10. PMID 33426938